CLINICAL TRIAL: NCT00803062
Title: A Randomized Phase III Trial of Cisplatin Plus Paclitaxel With and Without NCI-Supplied Bevacizumab (NSC #704865) Versus the Non-platinum Doublet, Topotecan Plus Paclitaxel, With and Without NCI-Supplied Bevacizumab, in Stage IVB, Recurrent or Persistent Carcinoma of the Cervix
Brief Title: Paclitaxel and Cisplatin or Topotecan With or Without Bevacizumab in Treating Patients With Stage IVB, Recurrent, or Persistent Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01084; NCI-2009-01084 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000628746; GOG-0240 (Other: NRG Oncology); GOG-0240 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Recurrent Cervical Carcinoma; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Paclitaxel; Taxes; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (paclitaxel and cisplatin) (Active Comparator): Patients receive paclitaxel IV over 3 hours or 24 hours on day 1 and cisplatin IV on day 1 or 2.
  Interventions: Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (paclitaxel, cisplatin, bevacizumab) (Experimental): Patients receive paclitaxel IV over 3 hours or 24 hours on day 1 and cisplatin IV and bevacizumab IV over 30-90 minutes on day 1 or 2.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (topotecan hydrochloride and paclitaxel) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1 and topotecan hydrochloride IV over 30 minutes on days 1-3.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Topotecan Hydrochloride
- Arm IV (topotecan hydrochloride, paclitaxel, bevacizumab) (Experimental): Patients receive paclitaxel IV over 3 hours and bevacizumab IV over 30-90 minutes on day 1 and topotecan hydrochloride IV over 30 minutes on days 1-3.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm II (paclitaxel, cisplatin, bevacizumab); Arm IV (topotecan hydrochloride, paclitaxel, bevacizumab)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm I (paclitaxel and cisplatin); Arm II (paclitaxel, cisplatin, bevacizumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Arm III (topotecan hydrochloride and paclitaxel); Arm IV (topotecan hydrochloride, paclitaxel, bevacizumab)

SUMMARY:
This randomized phase III trial studies the side effects of paclitaxel when given together with cisplatin or topotecan with or without bevacizumab and to compare how well they work in treating patients with stage IVB, cervical cancer that has come back or is persistent. Drugs used in chemotherapy, such as paclitaxel, cisplatin, and topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known whether paclitaxel is more effective when given together with cisplatin or topotecan with or without bevacizumab in treating patients with cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of bevacizumab to chemotherapy improves overall survival. Also to determine if a regimen involving paclitaxel and topotecan improves overall survival in comparison to a regimen involving cisplatin and paclitaxel. These regimens are to be evaluated in patients with stage IVB, recurrent, or persistent carcinoma of the cervix.

II. To determine and compare the frequency and severity of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 for the regimens administered on this study.

SECONDARY OBJECTIVES:

I. To estimate and compare the progression-free survival of patients treated by the regimens investigated on this study.

II. To estimate and compare the proportion of patients with tumor responses by the regimens investigated on this study.

TERTIARY OBJECTIVES:

I. To determine whether the addition of bevacizumab to chemotherapy, or the substitution of cisplatin with topotecan improve the health related quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy-Cervix Trial Outcome Index scale (FACT-Cx TOI) and produce favorable toxicity profiles (with a particular focus on peripheral neuropathy as measured by the Functional Assessment of Cancer Therapy-Gynecologic Oncology Group-Neurotoxicity version 4 [FACT/GOG-Ntx4] subscale and pain as measured by Brief Pain Inventory [BPI] single item).

II. To evaluate the impact of age, race, performance status, stage, histology, grade, disease site, prior chemotherapy with primary radiation, and time to recurrence on response rate, progression-free survival and overall survival of patients with metastatic/recurrent/persistent carcinoma of the cervix.

III. To determine the prevalence of active smoking in this cohort of recurrent cervical cancer patients.

IV. To estimate the extent of tobacco/nicotine dependence in the cohort. V. To determine if smoking is an independent risk factor for progression-free survival and overall survival in this population.

VI. To isolate, enumerate and characterize circulating tumor cells (CTC) recovered from blood drawn pre-cycle 1, pre-cycle 2 and pre-cycle 3 using the CTC-chip developed by the Massachusetts General Hospital (MGH) BioMEMS Resource Center and the MGH Cancer Center.

VII. To determine the association between CTC counts or characteristics and measures of clinical outcome.

VIII. To examine the association between angiogenesis markers in plasma (recovered from blood drawn pre-cycle 1, pre-cycle 2 and pre-cycle 3) and measures of clinical outcome.

IX. To evaluate the association between tumor markers of angiogenesis and hypoxia (using archival formalin-fixed and paraffin-embedded tumor tissue) and measures of clinical outcome.

X. To evaluate the association between single nucleotide polymorphisms (using deoxyribonucleic acid [DNA] extracted from whole blood) and measures of clinical outcome as well as measures of quality of life such as chemotherapy toxicity.

XI. To examine the relationship(s) among the various biomarkers. XII. To develop an optimal prognostic model for progression-free survival and overall survival using clinical covariates, smoking status and the various biomarkers.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours or 24 hours on day 1 and cisplatin IV on day 1 or 2.

ARM II: Patients receive paclitaxel IV over 3 hours or 24 hours on day 1 and cisplatin IV and bevacizumab IV over 30-90 minutes on day 1 or 2.

ARM III: Patients receive paclitaxel IV over 3 hours on day 1 and topotecan hydrochloride IV over 30 minutes on days 1-3.

ARM IV: Patients receive paclitaxel IV over 3 hours and bevacizumab IV over 30-90 minutes on day 1 and topotecan hydrochloride IV over 30 minutes on days 1-3.

In all arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have primary stage IVB, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy
* All patients must have measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT; biopsy confirmation is required if the lesion(s) measures < 30 mm or if the treating physician determines it is clinically indicated; patients must have at least one "target lesion" to be used to assess response on this protocol as defined by Response Evaluation Criteria in Solid Tumors (RECIST); this lesion should be the one that was biopsied if one was performed; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Absolute neutrophil count (ANC) >= 1500/mcl
* Platelets >= 100,000/mcl
* Serum creatinine =< upper limit of normal (ULN) (Common Toxicity Criteria [CTC] grade 0) or calculated creatinine clearance (Jeliffe formula) >= 60 ml/min
* Bilirubin =< 1.5 x institutional normal
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 x institutional normal
* Alkaline phosphatase =< 2.5 x institutional normal
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thrombo-embolus)
* Partial thromboplastin time (PTT) < 1.2 times the upper limit of normal
* Urine protein-creatinine ratio (UPC ratio) < 1.0
* Patients must have a GOG performance status of 0 or 1
* Patients must have recovered from the effects of surgery, radiation therapy, or chemoradiotherapy; at least six weeks must have elapsed from the last administration of chemoradiotherapy, and at least three weeks must have elapsed from the last administration of radiation therapy alone; at least six weeks must have elapsed from the time of any major surgical procedure prior to randomization
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet all of the pre-entry requirements, including baseline QOL questionnaire
* Patients must be free of active infection requiring antibiotics

Exclusion Criteria:

* Patients with bilateral hydronephrosis which cannot be alleviated by ureteral stents or percutaneous drainage
* Patients previously treated with chemotherapy except when used concurrently with radiation therapy

  * Patients who have received concurrent paclitaxel and/or concurrent topotecan with radiation therapy are ineligible
* Patients with craniospinal metastases
* Patients with a concomitant malignancy other than non-melanoma skin cancer
* Patients with a prior invasive malignancy (except non-melanoma skin cancer) who have had any evidence of disease within the last 5 years or whose prior malignancy treatment contraindicates the current protocol therapy
* Patients with serious non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess for which an interval of 3 to 6 months must pass before study entry; in addition, the patient must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation; patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg
  * Myocardial infarction or unstable angina < 6 months prior to registration
  * New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Serious cardiac arrhythmia requiring medication; this does not include asymptomatic, atrial fibrillation with controlled ventricular rate
  * CTCAE grade 2 or greater peripheral vascular disease (at least brief [< 24 hours (hrs)]) episodes of ischemia managed non-surgically and without permanent deficit)
  * History of CVA within six months
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients with or with anticipation of invasive procedures as defined below:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of bevacizumab therapy
  * Major surgical procedure anticipated during the course of the study; this includes, but is not limited to abdominal surgery (laparotomy or laparoscopy) prior to disease progression, such as colostomy or enterostomy reversal, interval or secondary cytoreductive surgery, or second look surgery; please consult with the study chair prior to patient entry for any questions related to the classification of surgical procedures
  * Core biopsy, within 7 days prior to randomization
* Patients who are pregnant or nursing; bevacizumab should not be administered to pregnant women; bevacizumab should not be administered to nursing women; patients of childbearing potential must agree to use contraceptive measures during study therapy and for at least six months after completion of bevacizumab therapy
* Patients who have received prior therapy with any anti-vascular endothelial growth factor (VEGF) drug, including bevacizumab
* Patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration and/or nutrition
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study; the investigator should feel free to consult the Study Chair or Study Co-Chairs for uncertainty in this regard
* Patients with significant peripheral vascular disease
* Patients with pre-existing grade 2 or greater peripheral neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2009-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krishnansu Tewari, Principal Investigator — NRG Oncology
Locations (549):
- United States (541):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Highlands Oncology Group PA - Fayetteville, Fayetteville, Arkansas
  - Washington Regional Medical Center - Fayetteville, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Roy and Patricia Disney Family Cancer Center, Burbank, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center - North Fresno, Fresno, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Advocate Lutheran General Hospital., Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Gynecologic Oncology of Indiana, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - Michiana Hematology Oncology-PC Westville, Westville, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - The Women's Institute for Gynecologic Cancer and Special Pelvic Surgery, Phillipsburg, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Queens Hospital Center, Jamaica, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System CCOP, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Saint Luke's Roosevelt Hospital Center - Saint Luke's Division, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Oncology Associates PA, Columbia, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Cancer Centers of the Carolinas-Greer Medical Oncology, Greer, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Tennessee Oncology PLLC- Centennial Medical Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University Medical Center Brackenridge, Austin, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Saint Luke's Episcopal Hospital, Houston, Texas
  - Veterans Administration Medical Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Fletcher Allen Health Care-Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Vince Lombardi Cancer Clinic, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Spain (8):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Gregorio Maranon, Madrid
  - M D Anderson International Spain, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Son Llatzer, Palma
  - Instituto Valenciano de Oncologia, Valencia

REFERENCES:
- [Derived] Tewari KS, Sill MW, Birrer MJ, Penson RT, Huang H, Moore DH, Ramondetta LM, Landrum LM, Oaknin A, Reid TJ, Leitao MM, Michael HE, Monk BJ. Final survival analysis of topotecan and paclitaxel for first-line treatment of advanced cervical cancer: An NRG oncology randomized study. Gynecol Oncol. 2023 Apr;171:141-150. doi: 10.1016/j.ygyno.2023.01.010. Epub 2023 Mar 8. PMID 36898292
- [Derived] Tewari KS, Sill MW, Monk BJ, Penson RT, Moore DH, Lankes HA, Ramondetta LM, Landrum LM, Randall LM, Oaknin A, Leitao MM, Eisenhauer EL, DiSilvestro P, Van Le L, Pearl ML, Burke JJ, Salani R, Richardson DL, Michael HE, Kindelberger DW, Birrer MJ. Circulating Tumor Cells In Advanced Cervical Cancer: NRG Oncology-Gynecologic Oncology Group Study 240 (NCT 00803062). Mol Cancer Ther. 2020 Nov;19(11):2363-2370. doi: 10.1158/1535-7163.MCT-20-0276. Epub 2020 Aug 26. PMID 32847980
- [Derived] Tewari KS, Sill MW, Penson RT, Huang H, Ramondetta LM, Landrum LM, Oaknin A, Reid TJ, Leitao MM, Michael HE, DiSaia PJ, Copeland LJ, Creasman WT, Stehman FB, Brady MF, Burger RA, Thigpen JT, Birrer MJ, Waggoner SE, Moore DH, Look KY, Koh WJ, Monk BJ. Bevacizumab for advanced cervical cancer: final overall survival and adverse event analysis of a randomised, controlled, open-label, phase 3 trial (Gynecologic Oncology Group 240). Lancet. 2017 Oct 7;390(10103):1654-1663. doi: 10.1016/S0140-6736(17)31607-0. Epub 2017 Jul 27. PMID 28756902
- [Derived] Penson RT, Huang HQ, Wenzel LB, Monk BJ, Stockman S, Long HJ 3rd, Ramondetta LM, Landrum LM, Oaknin A, Reid TJ, Leitao MM, Method M, Michael H, Tewari KS. Bevacizumab for advanced cervical cancer: patient-reported outcomes of a randomised, phase 3 trial (NRG Oncology-Gynecologic Oncology Group protocol 240). Lancet Oncol. 2015 Mar;16(3):301-11. doi: 10.1016/S1470-2045(15)70004-5. Epub 2015 Jan 29. PMID 25638326
- [Derived] Tewari KS, Sill MW, Long HJ 3rd, Penson RT, Huang H, Ramondetta LM, Landrum LM, Oaknin A, Reid TJ, Leitao MM, Michael HE, Monk BJ. Improved survival with bevacizumab in advanced cervical cancer. N Engl J Med. 2014 Feb 20;370(8):734-43. doi: 10.1056/NEJMoa1309748. PMID 24552320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 4/6/2009 and closed to accrual on 1/3/2012.
Groups:
- Arm I (Paclitaxel and Cisplatin): Paclitaxel 135 mg/m2 IV over 24 hrs on day 1 Cisplatin 50 mg/m2 IV on day 2 OR Paclitaxel 175 mg/m2 IV over 3 hrs on day 1 Cisplatin 50 mg/m2 IV on day 2 OR Paclitaxel 175 mg/m2 IV over 3 hrs on day 1 Cisplatin 50 mg/m2 IV on day 1 Cycles repeated q21 days to progression/toxicity
- Arm II (Paclitaxel, Cisplatin, Bevacizumab): Paclitaxel 135 mg/m2 IV over 24 hrs on day 1 Cisplatin 50 mg/m2 IV on day 2 Bevacizumab 15 mg/kg IV day 2 OR Paclitaxel 175 mg/m2 IV over 3 hrs on day 1 Cisplatin 50 mg/m2 IV on day 2 Bevacizumab 15 mg/kg IV day 2 OR Paclitaxel 175 mg/m2 IV over 3 hrs on day 1 Cisplatin 50 mg/m2 IV on day 1 Bevacizumab 15 mg/kg IV day 1 Cycles repeated q21 days to progression/toxicity
- Arm III (Topotecan Hydrochloride and Paclitaxel): Paclitaxel 175 mg/m2 over 3 hrs on day 1 Topotecan 0.75 mg/m2 over 30 mins days 1-3 Cycles repeated q21 days to progression/toxicity
- Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab): Paclitaxel 175 mg/m2 over 3 hrs on day 1 Topotecan 0.75 mg/m2 over 30 mins days 1-3 Bevacizumab 15 mg/kg IV day 1 Cycles repeated q21 days to progression/toxicity
Period: Overall Study
Arm/Group | Arm I (Paclitaxel and Cisplatin) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) | Arm III (Topotecan Hydrochloride and Paclitaxel) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab)
Started | 114 | 115 | 111 | 112
Completed | 114 | 115 | 111 | 112
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel and Cisplatin) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) | Arm III (Topotecan Hydrochloride and Paclitaxel) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab) | Total
Number analyzed (Participants) | 114 | 115 | 111 | 112 | 452
Age, Customized [Number; unit: participants]
  20-29 years | 6 | 5 | 1 | 6 | 18
  30-39 years | 25 | 27 | 30 | 12 | 94
  40-49 years | 36 | 34 | 33 | 41 | 144
  50-59 years | 27 | 28 | 24 | 37 | 116
  60-69 years | 14 | 13 | 17 | 12 | 56
  70-79 years | 5 | 5 | 5 | 4 | 19
  80-89 years | 1 | 3 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 115 | 111 | 112 | 452
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The observed length of life from randomization into the study to death or the date of last contact.
Time Frame: From entry into the study to death or the date of last contact, assessed up to 5 years
Population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel and Cisplatin) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) | Arm III (Topotecan Hydrochloride and Paclitaxel) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab)
Number analyzed (Participants) | 114 | 115 | 111 | 112
months | 14.26 [10.83 to 16.82] | 17.51 [13.96 to 22.93] | 12.68 [10.15 to 15.90] | 16.20 [12.71 to 18.96]

2. Primary Outcome: Progression-free Survival
Description: Disease that can be assessed clinically (physical examination) should be evaluated every cycle (every 3 weeks). Disease assessed by imaging modalities (CXR, CT, MRI) should be evaluated every other cycle unless other evidence of a change mandates earlier assessment. Tumor measurements should also be done after the final cycle (if the patient is taken off of study therapy for a reason other than progression) and then every 3 months x 2 years (followed with every 6 months x 3 years) until progression is documented. "Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions assessed radiographically and 50% increase if the only target lesion is a solitary pelvic mass measured by physical exam, or unequivocal progression of a non-target lesion, or the appearance of new lesions", or similar definition as accurate and appropriate.
Time Frame: From study entry until disease progression, death or date of last contact, assessed up to 5 years (During treatment: every 3 weeks if by physical exam, every 6 weeks by CXR, CT or MRI. In follow-up: quarterly for 2 years then semi-annually for 3 years)
Population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel and Cisplatin) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) | Arm III (Topotecan Hydrochloride and Paclitaxel) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab)
Number analyzed (Participants) | 114 | 115 | 111 | 112
months | 6.67 [5.72 to 8.08] | 9.63 [7.16 to 12.68] | 5.29 [4.27 to 6.80] | 7.36 [5.75 to 9.56]

3. Primary Outcome: Tumor Response
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions by CT, MRI or CXR. If the only target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% increase in longest diameter is required; Overall Response (OR) = CR + PR.
Time Frame: Every cycle (if assessed by physical exam), every other cycle (if assessed by imaging), after the final cycle, then every 3 months x 2 years, then every 6 months x 3 years up to 5 years.
Population: All randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Paclitaxel and Cisplatin) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) | Arm III (Topotecan Hydrochloride and Paclitaxel) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab)
Number analyzed (Participants) | 114 | 115 | 111 | 112
percentage of participants | 44.74 [35.42 to 54.34] | 49.57 [40.11 to 59.04] | 27.03 [19.03 to 36.28] | 47.32 [37.81 to 56.98]

4. Primary Outcome: To Determine and Compare the Frequency and Severity of Adverse Events as Assessed by CTCAE Version 3.0 for the Regimens Administered on This Study.
Description: The number of patients on each arm who have Grade 3 AE or higher toxicity.
Time Frame: From date of enrollment until 30 days after treatment completion
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel and Cisplatin) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) | Arm III (Topotecan Hydrochloride and Paclitaxel) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab)
Number analyzed (Participants) | 114 | 115 | 111 | 112
Participants
  Leukopenia | 34 | 48 | 48 | 66
  Thrombocytopenia | 6 | 5 | 5 | 9
  Neutropenia | 48 | 61 | 61 | 79
  Anemia | 33 | 29 | 23 | 30
  Other hematologic | 3 | 8 | 6 | 6
  Allergy/Immunology | 4 | 4 | 1 | 2
  Auditory/Ear | 1 | 1 | 0 | 0
  Cardiac | 2 | 16 | 4 | 14
  Coagulation | 4 | 4 | 1 | 0
  Constitutional | 12 | 16 | 13 | 16
  Dermatologic | 0 | 0 | 0 | 4
  Endocrine | 2 | 0 | 1 | 1
  Gastrointestinal | 22 | 29 | 11 | 22
  Genitourinary/Renal | 10 | 8 | 7 | 14
  Hemorrhage | 4 | 7 | 5 | 9
  Hepatobiliary | 0 | 0 | 0 | 1
  Infection | 17 | 18 | 19 | 30
  Lymphatics | 3 | 1 | 1 | 1
  Metabolic | 18 | 23 | 11 | 17
  Musculoskeletal | 0 | 2 | 2 | 2
  Neuropathy | 9 | 12 | 2 | 3
  Other Neurological | 8 | 5 | 7 | 9
  Pain | 21 | 30 | 22 | 27
  Pulmonary | 3 | 9 | 5 | 4
  Vascular | 8 | 17 | 6 | 7
  Death, Not CTC coded | 1 | 2 | 2 | 2

5. Other Pre Specified Outcome: Extent of Nicotine Dependence
Description: Assessed from answers the patients provide to a questionnaire. Will be assessed for associations with progression and/or death.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Health-related Quality of Life
Description: Assessed by FACT-Cx TOI; FACT/GOG-Ntx4 subscale; and BPI at baseline, before courses 2 and 5, and at 6 and 9 months after course 1. The linear mixed model will be used to evaluate the hypotheses on FACT-Cx TOI score, adjusting for baseline FACT-Cx TOI scores and age. A mixed-effects mixed-distribution model will be considered to analyze NTx4 subscale scores and the BPI score. 95% confidence intervals will be reported for the estimated treatment differences of BPI score.
Time Frame: Up to 9 months after course 1
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Levels of Angiogenesis Markers in Plasma
Description: Associations between biomarkers and overall survival or progression-free survival will be examined in a Cox proportional hazards model that includes significant prognostic variables based on prior research such as performance status, prior cisplatin therapy, and stage of disease. Logistic regression will be used to help assess the value of biomarkers in predicting response to a particular treatment or determine associations with response.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Levels of Cell-free DNA in Plasma
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Levels of Tumor Measures of Angiogenesis
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Number of CTCs
Description: as for outcome 7
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Prevalence of Active Smoking
Description: An estimate of the prevalence of active smoking will be calculated. Will be assessed for associations with progression and/or death.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment
Description: Adverse events number at risk reflects the number of patients who received treatment and submitted at least one adverse event form.
Arm/Group | Arm I (Paclitaxel and Cisplatin) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) | Arm III (Topotecan Hydrochloride and Paclitaxel) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 42/112 | 53/111 | 37/107 | 61/109
Other Adverse Events (participants affected / at risk) | 112/112 | 111/111 | 107/107 | 107/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel and Cisplatin) (N=112) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) (N=111) | Arm III (Topotecan Hydrochloride and Paclitaxel) (N=107) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab) (N=109)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Neutrophils (Blood and lymphatic system disorders) | 2 | 2 | 3 | 1
Platelets (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytes (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1
Vasovagal Episode (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 1 | 1 | 1
Hypertension (Cardiac disorders) | 0 | 2 | 0 | 1
Hypotension (Cardiac disorders) | 1 | 0 | 0 | 0
Inr (Vascular disorders) | 1 | 0 | 0 | 0
Dic (Vascular disorders) | 1 | 0 | 0 | 0
Fever (General disorders) | 1 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 2
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1 | 1 | 1 | 1
Death No Ctcae Term - Sudden Death (General disorders) | 0 | 0 | 0 | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Perforation, Gi - Colon (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fistula, Gi - Rectum (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Obstruction, Gi - Colon (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ulcer,gi - Rectum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Perforation, Gi - Rectum (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dental: Teeth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Leak, Gi - Rectum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Obstruction, Gi - Gallbladder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Anorexia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dehydration (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Perforation, Gi - Ileum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 1 | 2 | 1 | 3
Hemorrhage, Gu - Vagina (Vascular disorders) | 1 | 1 | 0 | 1
Hemorrhage/Pulmonary - Larynx (Vascular disorders) | 0 | 0 | 0 | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 0 | 0 | 1 | 1
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 0 | 0 | 0 | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 0 | 0 | 1 | 0
Hemorrhage, Gi - Esophagus (Vascular disorders) | 0 | 1 | 0 | 0
Hemorrhage, Gu - Ureter (Vascular disorders) | 0 | 0 | 0 | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 0 | 2 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 1 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 0 | 1 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 0 | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 0 | 0 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1 | 0 | 0 | 0
Febrile Neutropenia (Infections and infestations) | 3 | 1 | 5 | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 3 | 0 | 1 | 4
Inf Unknown Anc: Blood (Infections and infestations) | 0 | 1 | 0 | 1
Infection - Other (Infections and infestations) | 0 | 0 | 0 | 1
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Abdomen Nos (Infections and infestations) | 0 | 0 | 0 | 1
Inf Unknown Anc: Pelvis Nos (Infections and infestations) | 1 | 0 | 1 | 0
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 1 | 2 | 1 | 0
Inf Unknown Anc: Kidney (Infections and infestations) | 0 | 1 | 0 | 1
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 0 | 1 | 0 | 0
Inf Unknown Anc: Peritoneal Cavity (Infections and infestations) | 0 | 0 | 0 | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 0 | 0 | 2
Inf W/Gr 3 Or 4 Anc: Nerve-Peripheral (Infections and infestations) | 1 | 0 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 1 | 1 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 0 | 1 | 0 | 0
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Creatinine (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Muscle Weakness - Left-Sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Involuntary Movement (Nervous system disorders) | 0 | 1 | 0 | 0
Neurology - Other (Nervous system disorders) | 0 | 0 | 1 | 0
Mental Status (Nervous system disorders) | 0 | 1 | 0 | 0
Mood Alteration - Depression (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive Disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Pain - Other (General disorders) | 0 | 0 | 0 | 1
Pain: Pelvis (General disorders) | 0 | 3 | 1 | 0
Pain: Chest /Thorax Nos (General disorders) | 0 | 1 | 0 | 1
Pain: Pleura (General disorders) | 0 | 1 | 0 | 0
Pain: Neck (General disorders) | 0 | 1 | 0 | 0
Pain: Extremity-Limb (General disorders) | 1 | 2 | 0 | 1
Pain: Back (General disorders) | 2 | 1 | 0 | 1
Pain: Bone (General disorders) | 0 | 0 | 0 | 2
Pain: Rectum (General disorders) | 0 | 0 | 0 | 1
Pain: Abdominal Pain Nos (General disorders) | 4 | 4 | 2 | 6
Pain: Tumor (General disorders) | 0 | 1 | 0 | 0
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Ards (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 | 0 | 2 | 0
Stricture, Anastomotic, Gu - Ureter (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cystitis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 0 | 2 | 1
Fistula, Gu - Vagina (Renal and urinary disorders) | 2 | 2 | 0 | 2
Fistula, Gu - Genital Tract-Female (Renal and urinary disorders) | 0 | 0 | 1 | 1
Fistula, Gu - Bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 3 | 0 | 0 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 7 | 8 | 3 | 3
Death No Ctcae Term - Multi-Organ Failure (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel and Cisplatin) (N=112) | Arm II (Paclitaxel, Cisplatin, Bevacizumab) (N=111) | Arm III (Topotecan Hydrochloride and Paclitaxel) (N=107) | Arm IV (Topotecan Hydrochloride, Paclitaxel, Bevacizumab) (N=109)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 19 | 20 | 5 | 4
Rhinitis (Immune system disorders) | 6 | 11 | 5 | 10
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 | 1 | 0 | 1
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1 | 3 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 17 | 7 | 3 | 5
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Neutrophils (Blood and lymphatic system disorders) | 79 | 90 | 75 | 93
Platelets (Blood and lymphatic system disorders) | 39 | 55 | 45 | 61
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 | 2 | 2 | 3
Leukocytes (Blood and lymphatic system disorders) | 88 | 95 | 89 | 99
Lymphopenia (Blood and lymphatic system disorders) | 4 | 12 | 8 | 13
Hemoglobin (Blood and lymphatic system disorders) | 107 | 101 | 104 | 101
Palpitations (Cardiac disorders) | 2 | 3 | 3 | 1
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 3 | 2 | 0 | 1
Vasovagal Episode (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Hypertension (Cardiac disorders) | 10 | 36 | 3 | 27
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac General - Other (Cardiac disorders) | 2 | 0 | 0 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 3 | 3 | 3 | 2
Inr (Vascular disorders) | 4 | 5 | 1 | 0
Coagulopathy - Other (Vascular disorders) | 0 | 0 | 0 | 1
Ptt (Vascular disorders) | 1 | 6 | 0 | 3
Constitutional Symptoms - Other (General disorders) | 2 | 1 | 2 | 1
Sweating (General disorders) | 9 | 3 | 5 | 4
Weight Gain (General disorders) | 3 | 5 | 6 | 9
Patient Odor (General disorders) | 0 | 0 | 0 | 1
Fever (General disorders) | 16 | 17 | 13 | 16
Weight Loss (General disorders) | 9 | 26 | 6 | 19
Rigors/Chills (General disorders) | 7 | 3 | 3 | 5
Fatigue (General disorders) | 93 | 91 | 76 | 82
Insomnia (General disorders) | 18 | 15 | 15 | 28
Nail Changes (Skin and subcutaneous tissue disorders) | 2 | 5 | 3 | 6
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 69 | 65 | 69 | 71
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Bruising (Skin and subcutaneous tissue disorders) | 4 | 3 | 4 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 14 | 13 | 16 | 18
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 4 | 6 | 4
Decubitus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 6 | 5 | 5
Burn (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Flushing (Skin and subcutaneous tissue disorders) | 5 | 3 | 4 | 2
Hand-Foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 5 | 7 | 4 | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 7 | 0 | 3
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Hot Flashes (Endocrine disorders) | 14 | 12 | 11 | 13
Diabetes (Endocrine disorders) | 0 | 1 | 1 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 1 | 0
Endocrine - Other (Endocrine disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 1
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Ulcer,gi - Anus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary Gland Changes (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Ulcer,gi - Esophagus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental: Periodontal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fistula, Gi - Rectum (Gastrointestinal disorders) | 0 | 5 | 0 | 4
Obstruction, Gi - Colon (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 3 | 0 | 3
Esophagitis (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 7 | 1 | 3
Ulcer,gi - Rectum (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Heartburn (Gastrointestinal disorders) | 7 | 18 | 8 | 4
Mucositis (Functional/Sympt) - Esophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental: Teeth (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Mucositis (Functional/Sympt) - Pharynx (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 3 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 5 | 0 | 1
Distention (Gastrointestinal disorders) | 1 | 5 | 2 | 0
Taste Alteration (Gastrointestinal disorders) | 10 | 11 | 9 | 13
Incontinence, Anal (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 3 | 2 | 5
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 7 | 6 | 3 | 10
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Mucositis (Clinical Exam) - Rectum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Obstruction, Gi - Jejunum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dentures (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 7 | 7 | 8 | 10
Vomiting (Gastrointestinal disorders) | 37 | 47 | 30 | 28
Anorexia (Gastrointestinal disorders) | 30 | 42 | 27 | 33
Dehydration (Gastrointestinal disorders) | 6 | 12 | 4 | 3
Constipation (Gastrointestinal disorders) | 62 | 54 | 49 | 52
Nausea (Gastrointestinal disorders) | 77 | 75 | 56 | 63
Gastrointestinal - Other (Gastrointestinal disorders) | 3 | 4 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 38 | 46 | 39 | 35
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 6 | 7 | 3 | 8
Hemorrhage, Gu - Vagina (Vascular disorders) | 16 | 14 | 10 | 10
Hemorrhage, Gu - Urethra (Vascular disorders) | 0 | 0 | 0 | 1
Hemorrhage/Pulmonary - Lung (Vascular disorders) | 0 | 0 | 0 | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 3 | 8 | 6 | 10
Hemorrhage/Pulmonary - Respiratory Tract Nos (Vascular disorders) | 0 | 0 | 1 | 0
Hemorrhage, Gi - Varices (Rectal) (Vascular disorders) | 0 | 1 | 0 | 0
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1 | 15 | 2 | 22
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hemorrhage, Gi - Anus (Vascular disorders) | 1 | 1 | 0 | 2
Hemorrhage, Gu - Ureter (Vascular disorders) | 1 | 1 | 1 | 1
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 0 | 3 | 0 | 7
Hemorrhage, Gu - Kidney (Vascular disorders) | 0 | 1 | 0 | 0
Hemorrhage, Gu - Bladder (Vascular disorders) | 0 | 5 | 1 | 2
Hemorrhage, Gi - Colon (Vascular disorders) | 0 | 0 | 0 | 1
Hemorrhage, Cns (Vascular disorders) | 0 | 1 | 0 | 0
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 | 1 | 0 | 1
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pancreatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 0 | 1 | 0 | 2
Inf W/Gr 3 Or 4 Anc: Dental-Tooth (Infections and infestations) | 0 | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: External Ear (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 0 | 0 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 0 | 5 | 3 | 4
Inf W/Gr 3 Or 4 Anc: Lip/Perioral (Infections and infestations) | 1 | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 1 | 1 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Joint (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1 | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1 | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 1 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Otitis Media Nos (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 2 | 4 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1 | 0 | 0 | 0
Febrile Neutropenia (Infections and infestations) | 4 | 2 | 2 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Lip/Perioral (Infections and infestations) | 0 | 0 | 0 | 2
Inf Unknown Anc: Nerve-Peripheral (Infections and infestations) | 0 | 0 | 0 | 1
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 0 | 1 | 2
Inf Unknown Anc: Sinus (Infections and infestations) | 2 | 0 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 0 | 0 | 0 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 0 | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 7 | 17 | 11 | 15
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 0 | 2 | 0 | 0
Infection - Other (Infections and infestations) | 3 | 6 | 6 | 6
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 0 | 2 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Nerve-Peripheral (Infections and infestations) | 1 | 0 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Conjunctiva (Infections and infestations) | 0 | 0 | 1 | 0
Inf Unknown Anc: Vagina (Infections and infestations) | 0 | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Mucosa (Infections and infestations) | 0 | 1 | 0 | 0
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 0 | 1 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 0 | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 0 | 0 | 4 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 1 | 0 | 1 | 3
Inf Unknown Anc: Bronchus (Infections and infestations) | 0 | 0 | 1 | 1
Inf Unknown Anc: Eye Nos (Infections and infestations) | 0 | 0 | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 3 | 6 | 7 | 8
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 0 | 0 | 2 | 1
Inf Unknown Anc: Wound (Infections and infestations) | 1 | 0 | 0 | 0
Inf Unknown Anc: Dental-Tooth (Infections and infestations) | 0 | 2 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Vulva (Infections and infestations) | 0 | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Pelvis Nos (Infections and infestations) | 0 | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 0 | 0 | 2 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Anal/Perianal (Infections and infestations) | 0 | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Sinus (Infections and infestations) | 1 | 0 | 1 | 2
Inf W/Gr 3 Or 4 Anc: Pharynx (Infections and infestations) | 0 | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Bronchus (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Ureter (Infections and infestations) | 0 | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Lymphatic (Infections and infestations) | 0 | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2 | 4 | 1 | 1
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 2 | 3 | 6 | 4
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 0 | 1 | 0 | 1
Lymphatics - Other (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1
Edema: Limb (Blood and lymphatic system disorders) | 26 | 15 | 23 | 19
Edema: Head And Neck (Blood and lymphatic system disorders) | 2 | 1 | 2 | 1
Dermal Change (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Ast (Metabolism and nutrition disorders) | 6 | 17 | 9 | 7
Gfr (Metabolism and nutrition disorders) | 1 | 3 | 3 | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 5 | 3 | 6 | 4
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Proteinuria (Metabolism and nutrition disorders) | 4 | 16 | 3 | 7
Hemoglobinuria (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Creatinine (Metabolism and nutrition disorders) | 16 | 24 | 6 | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 | 19 | 11 | 16
Ggt (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Alt (Metabolism and nutrition disorders) | 7 | 15 | 5 | 5
Alkaline Phosphatase (Metabolism and nutrition disorders) | 15 | 21 | 11 | 11
Bilirubin (Metabolism and nutrition disorders) | 3 | 4 | 1 | 2
Lipase (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 4 | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 8 | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 11 | 24 | 10 | 17
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 2 | 6 | 1 | 1
Amylase (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 21 | 7 | 11
Hyperkalemia (Metabolism and nutrition disorders) | 8 | 9 | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 24 | 27 | 19 | 29
Hypokalemia (Metabolism and nutrition disorders) | 18 | 24 | 12 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 5 | 1 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 3 | 4 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 29 | 40 | 6 | 13
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1
Joint-Function (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Extremity-Upper (Function) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Gait/Walking (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 14 | 12 | 7 | 15
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 3 | 7 | 3 | 3
Syncope (Nervous system disorders) | 2 | 1 | 3 | 4
Involuntary Movement (Nervous system disorders) | 0 | 1 | 0 | 2
Psychosis (Nervous system disorders) | 0 | 1 | 0 | 0
Neurology - Other (Nervous system disorders) | 4 | 1 | 0 | 3
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 19 | 16 | 14 | 13
Mood Alteration - Anxiety (Nervous system disorders) | 14 | 20 | 9 | 16
Mood Alteration - Agitation (Nervous system disorders) | 2 | 3 | 1 | 1
Tremor (Nervous system disorders) | 1 | 2 | 1 | 1
Speech Impairment (Nervous system disorders) | 0 | 0 | 0 | 2
Seizure (Nervous system disorders) | 1 | 1 | 0 | 0
Personality (Nervous system disorders) | 1 | 0 | 0 | 0
Irritability (Nervous system disorders) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive Disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 2 | 3 | 1
Confusion (Nervous system disorders) | 3 | 4 | 0 | 1
Memory Impairment (Nervous system disorders) | 2 | 2 | 3 | 5
Dizziness (Nervous system disorders) | 13 | 9 | 10 | 11
Neuropathy,cranial - Cn Viii Hearing/Balance (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy,cranial - Cn Ii Vision (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy,cranial - Cn I Smell (Nervous system disorders) | 0 | 2 | 0 | 0
Neuropathy-Sensory (Nervous system disorders) | 76 | 64 | 63 | 71
Neuropathy-Motor (Nervous system disorders) | 7 | 2 | 4 | 4
Ocular/Visual - Other (Eye disorders) | 1 | 0 | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 0 | 0 | 0
Watery Eye (Eye disorders) | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 2
Ocular Surface Disease (Eye disorders) | 1 | 0 | 0 | 0
Flashing Lights/Floaters (Eye disorders) | 2 | 1 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Blurred Vision (Eye disorders) | 10 | 7 | 4 | 10
Pain - Other (General disorders) | 7 | 12 | 11 | 6
Pain: Urethra (General disorders) | 0 | 3 | 0 | 3
Pain: Perineum (General disorders) | 0 | 2 | 1 | 1
Pain: Pelvis (General disorders) | 8 | 15 | 11 | 13
Pain: Breast (General disorders) | 2 | 0 | 0 | 0
Pain: Vagina (General disorders) | 3 | 5 | 2 | 2
Pain: Chest /Thorax Nos (General disorders) | 7 | 3 | 6 | 3
Pain: Chest Wall (General disorders) | 2 | 4 | 2 | 5
Pain: Throat/Pharynx/Larynx (General disorders) | 2 | 1 | 4 | 6
Pain: Pleura (General disorders) | 0 | 0 | 1 | 0
Pain: Head/Headache (General disorders) | 12 | 26 | 17 | 21
Pain: Neck (General disorders) | 0 | 5 | 1 | 1
Pain: Extremity-Limb (General disorders) | 26 | 18 | 18 | 18
Pain: Buttock (General disorders) | 3 | 3 | 0 | 3
Pain: Back (General disorders) | 25 | 23 | 16 | 22
Pain: Joint (General disorders) | 17 | 24 | 23 | 24
Pain: Bone (General disorders) | 7 | 12 | 15 | 9
Pain: Kidney (General disorders) | 2 | 0 | 1 | 1
Pain: Bladder (General disorders) | 5 | 2 | 3 | 3
Pain: Pain Nos (General disorders) | 4 | 8 | 3 | 4
Pain: Stomach (General disorders) | 1 | 2 | 0 | 1
Pain: Rectum (General disorders) | 2 | 6 | 1 | 8
Pain: Peritoneum (General disorders) | 0 | 1 | 0 | 0
Pain: Oral Cavity (General disorders) | 0 | 3 | 0 | 1
Pain: Dental/Teeth/Peridontal (General disorders) | 2 | 2 | 1 | 0
Pain: Abdominal Pain Nos (General disorders) | 41 | 38 | 30 | 33
Pain: Scalp (General disorders) | 0 | 1 | 0 | 0
Pain: Oral - Gums (General disorders) | 1 | 0 | 1 | 0
Pain: Skin (General disorders) | 1 | 0 | 2 | 0
Pain: Middle Ear (General disorders) | 1 | 3 | 0 | 1
Pain: External Ear (General disorders) | 0 | 1 | 0 | 0
Pain: Cardiac/ Heart (General disorders) | 1 | 0 | 0 | 0
Pain: Tumor (General disorders) | 2 | 1 | 0 | 1
Pain: Muscle (General disorders) | 21 | 17 | 21 | 25
Pain: Neuralgia (General disorders) | 2 | 1 | 3 | 0
Pain: Sinus (General disorders) | 0 | 1 | 1 | 3
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 2
Airway Obstruction - Bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 10
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 1 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 12 | 24 | 21
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 29 | 26 | 22 | 23
Renal/Genitourinary - Other (Renal and urinary disorders) | 3 | 6 | 5 | 4
Leak, Gu - Vagina (Renal and urinary disorders) | 1 | 0 | 0 | 1
Leak, Gu - Urethra (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cystitis (Renal and urinary disorders) | 0 | 3 | 3 | 3
Urinary Color Change (Renal and urinary disorders) | 1 | 2 | 3 | 2
Urinary Retention (Renal and urinary disorders) | 2 | 4 | 4 | 0
Urinary Electrolyte Wasting (Renal and urinary disorders) | 1 | 0 | 1 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 2 | 4 | 4 | 3
Incontinence, Urinary (Renal and urinary disorders) | 9 | 7 | 9 | 8
Fistula, Gu - Vagina (Renal and urinary disorders) | 3 | 1 | 1 | 1
Fistula, Gu - Bladder (Renal and urinary disorders) | 0 | 1 | 0 | 1
Bladder Spasm (Renal and urinary disorders) | 0 | 4 | 2 | 2
Renal Failure (Renal and urinary disorders) | 1 | 1 | 0 | 2
Urinary Frequency (Renal and urinary disorders) | 10 | 11 | 7 | 8
Libido (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Irregular Menses (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Vaginitis (Reproductive system and breast disorders) | 2 | 1 | 0 | 1
Vaginal Stenosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 7 | 5 | 10 | 9
Syndromes - Other (General disorders) | 1 | 0 | 2 | 0
Cytokine Release Syndrome (General disorders) | 1 | 1 | 0 | 0
Flu-Like Syndrome (General disorders) | 0 | 4 | 1 | 1
Vascular - Other (Vascular disorders) | 1 | 0 | 0 | 0
Vein Injury - Other Nos (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1 | 1 | 0 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 | 12 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less